CLINICAL TRIAL: NCT05693532
Title: Probing the Rheumatoid Arthritis Brain to Elucidate Central Pain Pathways
Acronym: Pro-BEPP
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN19RH007
Record Dates: First submitted 2022-12-21; First posted 2023-01-23 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples will be taken for peripheral immunophenotyping including proteomic and transcriptomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rheumatoid arthritis (RA) is a common disease which is characterised by severe joint inflammation and chronic pain. The discovery of new joint specific treatments has transformed patient outcomes and yet most patients, even those whose joints respond fully to these treatments, continue to experience significant levels of pain. The investigators therefore believe that RA pain is caused by alternative sources in addition to the joints. Our group are pioneering the investigation of a possible link between the brain and the pain which RA patients experience. By employing sophisticated brain scanning methods, the investigators have shown that high levels of pain and blood inflammation are associated with changes within a specific region of the brain known as the left inferior parietal lobule(L-IPL). This region exhibited abnormal connections with other brain regions already known to be associated with pain in another chronic pain disorder called fibromyalgia. Fibromyalgia is a musculoskeletal condition which is not classically related to high levels of blood inflammation, although, interestingly, it is not uncommon for it to co-exist in RA patients. In light of our preliminary brain scan studies, the investigators now think that fibromyalgia in the context of RA may be partially influenced by inflammation. In order to fully understand the precise processes that lead to this potential relationship, it is important to characterise the biological abnormalities that underlie our brain scan observations. Previous animal experiments have consistently observed abnormalities, such as high levels of the brain chemical glutamate and haphazard brain activity, in the context of inflammation. Conducting similar experiments in humans is not practical due to the inherent dangers of sampling live brain tissue. Instead, neuroscientists commonly use non-invasive methods to manipulate specific parts of the brain in order to better understand how they function. In conjunction, the latest scanners are now able to indirectly measure the effect of the brain modulation on relevant aspects of brain biology without the need to remove tissue. This information will help us to better understand the relationship between inflammation and pain in the RA brain.

DETAILED DESCRIPTION:
Rheumatoid Arthritis-related pain is only partially explained by joint specific inflammation. Despite excellent control of peripheral inflammation by contemporary immune modulatory regimes, as many as 50% of patients continue to report disabling levels of pain, thus comprising an urgent unmet clinical need. The investigators have been among the first to evidence a contributory role of the central nervous system (CNS) as an explanation for this apparent disconnect. Our cross-sectional neuroimaging studies have implicated the left inferior parietal lobule of the brain as a critical interface between inflammation and pain. Not only did this region associate with levels of patient reported pain and indicators of systemic inflammation, but it was found to be functionally hyperconnected to brain networks established to be pro-nociceptive in CNS based chronic pain disorders such as fibromyalgia. In parallel, preclinical experiments suggest that systemic inflammation leads to heightened glutamate neurotransmission, which in turn results in disorganised neuronal signal activity and ultimately altered functional connectivity between regions of the brain. In RA patients, the investigators hypothesise that systemic inflammation-related neural glutamate enhancement triggers chaotic neuronal signaling, followed by compensatory hyperconnectivity with pro-nociceptive functional brain networks. Thereby, the investigators believe that dysfunctional inflammatory processes in RA not only mediate nociception in vulnerable joints but also nociception in vulnerable regions of the brain.

Given the clear practical constraints of sampling fresh human brain tissue, the investigators propose to test our hypothesis by combining state-of-the-art non-invasive brain modulatory techniques alongside leading-edge neurobiological surrogate imaging measures. Transcranial magnetic stimulation (TMS) is the neural modulatory probe of choice for neuroscientists seeking to infer causality of specific brain cortical regions. Ultra-high resolution 7T MRI enables measurement of functional connectivity and haphazard neuronal signal activity at significantly superior spatial resolution compared to standard 3T approaches and can uniquely assess regional glutamate. As a critical first step, this feasibility study aims to pilot a transcranial magnetic stimulation (TMS) protocol designed to target the L-IPL in RA. The investigators will evaluate its effect employing ultra-high resolution 7T functional and glutamate measures. This novel project will inform a larger study which will aim to provide more robust evidence for the proposed neural pain interface between systemic inflammation and pain. Such knowledge could potentially support the analgesic testing of existing compounds e.g. alternative/augmented immunosuppressants or neural glutamate modulatory agents; and reverse translated in order to more precisely dissect the culprit mechanisms which in turn may inform the development of novel pain therapeutics. Both represent core aims of Versus Arthritis and address critical priorities among the patient populations that the investigators serve.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years < 75 years.
* Physician diagnosis of RA
* ACR definition of chronic widespread pain
* Able and willing to maintain usual/ medication for the 6-week study duration
* CRP > 6mg/L or ESR > 20mm/hr

  •≥1 swollen joint
* Right-handed (to reduce neuroimaging heterogeneity)

Exclusion Criteria:

* Inability to provide written informed consent.
* Severe physical impairment (e.g. blindness, deafness, paraplegia).
* Pregnant, planning pregnancy or breast feeding.
* Severe claustrophobia precluding MRI.
* Contraindications to MRI(e.g. metal implants/ pacemaker).
* Contraindication to TMS (e.g. history of seizures).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve participants aged over 18 years with active inflammatory RA who meet the inclusion criteria below and who have none of the specified exclusion criteria. All will give full informed consent. Rheumatoid arthritis patients attending secondary care clinics in NHS GG&C and in NHS Lanarkshire will be screened for eligibility. NHS Lanarkshire will act as a participant identification centre (PIC) and all study participants will undertake study procedures at the University of Glasgow and the Queen Elizabeth University Hospital (NHS GG&C).
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Changes in functional connectivity and neuronal signal cohesion | 2 hours
  Changes in functional connectivity and neuronal signal cohesion as measured by 7T MRI. Changes are baseline to post-treatment/sham.
Changes in glutamate signal | 2 hours
  Changes in glutamate signal in the L-IPL as measured by 7T MRS . Changes are baseline to post-treatment/sham.

SECONDARY OUTCOMES:
Changes in pain severity | 2 weeks
  Changes in global pain as measures by the Pain-NRS scale from baseline to 2-hours post-treatment/sham and from baseline to 2-week follow up.
Changes from the Michigan Body Map Regional Pain. | 2 weeks
  Changes in regional pain severity as measured by the Michigan Body Map Regional Pain from baseline to 2-week follow-up.
Changes in RA disease activity as measured by SDAI. | 2 weeks
  Changes in Rheumatoid Arthritis disease activity as measured by the Simplified Disease Activity Index (SDAI) from baseline to 2-hours post-treatment/sham and from baseline to 2-week follow up.
Changes in RA disease activity as measured by CDAI. | 2 weeks
  Changes in Rheumatoid Arthritis disease activity as measured by the Clinical Disease Activity Index (CDAI) from baseline to 2-hours post-treatment/sham and from baseline to 2-week follow up.
Changes in putative pain confounders as measured by PROMIS-Fatigue | 2 weeks
  Changes in putative pain confounders as measured by PROMIS-Fatigue from baseline to 2-week follow-up.
  PROMIS stands for 'Patient-Reported Outcomes Measurement Information System'. Measures are scored via T-score metric where 50 is the mean of a relevant reference population and 10 is the standard deviation.
  On the T-score metric:
  * A score of 40 is one standard deviation lower than the mean of the reference population.
  * A score of 60 is one standard deviation higher than the mean of the reference population.
  The lower score indicates less of the concept being measured; the higher score indicates more of the concept being measured.
Changes in putative pain confounders as measured by PROMIS-Depression | 2 weeks
  Changes in putative pain confounders as measured by PROMIS-Depression, from baseline to 2-week follow-up.
  PROMIS stands for 'Patient-Reported Outcomes Measurement Information System'. Measures are scored via T-score metric where 50 is the mean of a relevant reference population and 10 is the standard deviation.
  On the T-score metric:
  * A score of 40 is one standard deviation lower than the mean of the reference population.
  * A score of 60 is one standard deviation higher than the mean of the reference population.
  The lower score indicates less of the concept being measured; the higher score indicates more of the concept being measured.
Changes in putative pain confounders as measured by PROMIS-Anxiety | 2 weeks
  Changes in putative pain confounders as measured by PROMIS-Anxiety from baseline to 2-week follow-up.
  PROMIS stands for 'Patient-Reported Outcomes Measurement Information System'. Measures are scored via T-score metric where 50 is the mean of a relevant reference population and 10 is the standard deviation.
  On the T-score metric:
  * A score of 40 is one standard deviation lower than the mean of the reference population.
  * A score of 60 is one standard deviation higher than the mean of the reference population.
  The lower score indicates less of the concept being measured; the higher score indicates more of the concept being measured.
Changes in putative pain confounders as measured by PROMIS-Sleep Related Impairment | 2 weeks
  Changes in putative pain confounders as measured by PROMIS-Sleep Related Impairment, from baseline to 2-week follow-up.
  PROMIS stands for 'Patient-Reported Outcomes Measurement Information System'. Measures are scored via T-score metric where 50 is the mean of a relevant reference population and 10 is the standard deviation.
  On the T-score metric:
  * A score of 40 is one standard deviation lower than the mean of the reference population.
  * A score of 60 is one standard deviation higher than the mean of the reference population.
  The lower score indicates less of the concept being measured; the higher score indicates more of the concept being measured.
Changes in putative pain confounders as measured by PROMIS-Physical functioning short form | 2 weeks
  Changes in putative pain confounders as measured by PROMIS-Physical functioning short form from baseline to 2-week follow-up.
  PROMIS stands for 'Patient-Reported Outcomes Measurement Information System'. Measures are scored via T-score metric where 50 is the mean of a relevant reference population and 10 is the standard deviation.
  On the T-score metric:
  * A score of 40 is one standard deviation lower than the mean of the reference population.
  * A score of 60 is one standard deviation higher than the mean of the reference population.
  The lower score indicates less of the concept being measured; the higher score indicates more of the concept being measured.
Changes in putative pain confounders as measured by PROMIS-Pain Interference | 2 weeks
  Changes in putative pain confounders as measured by PROMIS-Pain Interference from baseline to 2-week follow-up.
  PROMIS stands for 'Patient-Reported Outcomes Measurement Information System'. Measures are scored via T-score metric where 50 is the mean of a relevant reference population and 10 is the standard deviation.
  On the T-score metric:
  * A score of 40 is one standard deviation lower than the mean of the reference population.
  * A score of 60 is one standard deviation higher than the mean of the reference population.
  The lower score indicates less of the concept being measured; the higher score indicates more of the concept being measured.
Changes in putative pain confounders as measured by ACR Fibromyalgia Scale | 2 weeks
  Changes in putative pain confounders as measured by ACR Fibromyalgia Scale from baseline to 2-week follow-up.
Changes in blood protein levels of inflammatory cytokines/chemokines. | 2 weeks
  Changes in blood protein levels of inflammatory cytokines/chemokines from baseline to 2-week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Basu, MD, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, Scotland, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT05693532/Prot_000.pdf